CLINICAL TRIAL: NCT05362591
Title: Biomimetic Anterior Resin Bonded Restorations for Adolescent Patients
Brief Title: Anterior Resin Bonded Restorations for Adolescent
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Naglaa Ibrahim Ezz, Associate professor, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-D124-2
Record Dates: First submitted 2022-04-23; First posted 2022-05-05 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Missing Teeth
Keywords: missing incisors; resin bonded bridge
MeSH Terms: conditions — Anodontia | interventions — Denture, Partial, Fixed, Resin-Bonded

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resin bonded bridge with no preparation (Experimental): resin bonded bridge without enamel preparation
  Interventions: Procedure: resin bonded bridge with no preparation
- resin bonded bridge with minimal preparation (Active Comparator): resin bonded bridge with minimal preparation on tooth enamel
  Interventions: Procedure: resin bonded bridge with minimal preparation

INTERVENTIONS:
Procedure: resin bonded bridge with no preparation — resin bonded bridge without enamel preparation
  Arms: resin bonded bridge with no preparation
Procedure: resin bonded bridge with minimal preparation — resin bonded bridge with minimal preparation of tooth enamel
  Arms: resin bonded bridge with minimal preparation

SUMMARY:
a 24 Patients above 12 years old with missing upper incisor were divided into two groups, group 1: 12 patient will be treated by resin bonded bridge (RBB) with no preparation protocol, group 2: 12 patient will be treated by resin bonded bridge (RBB) with minimal preparation protocol.

(RBB) retention/survival, patient's speech as well as thermal sensitivity and patient's satisfaction will be evaluated for 12 month at 3,6,9 and 12 month.

ELIGIBILITY:
Inclusion Criteria:

1. 12-18 years old
2. Full set of permanent teeth.
3. Missing upper incisor
4. Controlled dental disease - no active caries or periodontal diseases
5. Patients will be available to be clinically reviewed up to 1 year

Exclusion Criteria:

1. Patients with uncontrolled active tooth decay or periodontal disease (i.e. 4+ mm probing depth and bleeding on probing).
2. Patients with teeth missing opposite to the planned RBB
3. Abutment tooth mobility of 2 or greater (Millers classification)
4. Patients with debilitating illnesses or complicating medical conditions
5. Heavily restored tooth abutment not suitable for an RBB

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-05-08 (Actual); Primary Completion 2024-05-04 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
resin bonded bridge retention/survival | 12 month
  Presence of the prosthesis in patient's mouth (Yes/No) by clinical visual examination.

SECONDARY OUTCOMES:
Patient's satisfaction | 12 month
  Patient satisfaction outcome is including the following: comfort and stability, esthetics, ease of cleaning, ability to speak, self-esteem, and functionality. the outcome will be evaluated by a visual analogue scale ranging from 0 to 10, where 10 is the maximum (better outcome) and 0 is the minimum (worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- October university for modern sciences and arts, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided